CLINICAL TRIAL: NCT06808334
Title: CLAiR Pivotal Study
Status: Recruiting | Type: Observational
Sponsor: Toku Eyes Ltd (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CPS-En01
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: No Condition
Keywords: retinal image; ASCVD; AI; cardiovascular risk; adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Other: CLAIR — Subject will have retinal images obtained and uploaded to CLAiR Software. Subjects are not directly in contact with CLAiR software. There is no medical intervention.

SUMMARY:
This is a multi-site, observational clinical study to validate the performance of the CLAiR AI software in identifying elevated atherosclerotic cardiovascular disease (ASCVD) risk from retinal (eye) images obtained from two different retinal image camera models.

DETAILED DESCRIPTION:
This is a prospective observational clinical study to collect retinal images and clinical biomarker data in order to analyze the performance of the CLAiR SaMD compared to the reference PCE risk score. CLAiR is a deep learning (DL) model that uses retinal photographs and limited demographic data to classify an individual's risk of developing ASCVD over the next 10 years as elevated (≥7.5%) or non-elevated (<7.5%). For validation, the output of the algorithm can be directly compared to the PCE output, a widely accepted algorithm used by Healthcare Providers to predict ASCVD risk in patients.

The primary hypothesis is that the CLAiR SaMD can achieve high sensitivity and specificity in the binary determination of Yes/No elevated ASCVD risk with PCE risk score ≥7.5% as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 40-75 years
2. Participants must be capable of providing informed consent, demonstrating understanding of the study details, and willingly sign a consent form or verbally confirm their consent in the presence of a witness.
3. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known history of atherosclerotic cardiovascular disease, including stroke, heart attack, coronary artery surgery, or stenting
2. Current use of cholesterol-lowering medication, such as a statin
3. Pregnancy
4. A person who has (in at least one eye):

   * Persistent vision impairment: legally blind when wearing current driving glasses or known VA<20/400
   * Known pathological myopia
   * Previous treatment or currently under the care for a retinal disease by a specialist (e.g., ophthalmologist)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and Females between the ages of 40-75 years of age.
Sampling Method: Probability Sample
Enrollment: 942 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that CLAiR can accurately identify elevated ASCVD risk as determined by PCE score. | through study completion, an average of 6 months
  Sensitivity and Specificity of CLAiR binary elevated risk classification (PCE ≥ 7.5% Y/N) against the reference standard of PCE ≥ 7.5%

CONTACTS AND LOCATIONS:
Overall Officials: Michael McConnell, MD, Study Director — Toku Inc.
Locations (1):
- Diabetes and Endocrine Associates of Stark County, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No